CLINICAL TRIAL: NCT06391905
Title: PCSK9 Inhibitors in Combination With Advanced Treatment Strategies for the Treatment of Advanced Colorectal Cancer With pMMR/MSS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yong Li, MD, Chief Physician of Gastrointestinal Surgery, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lron-Man 02
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: pMMR/MSS; PCSK9; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Experimental: Advanced Treatment combined with PCSK9 inhibitor Control: Advanced Treatmentcombined without PCSK9 inhibitor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Late standard first-line treatment regimen group (Other): Fluorouracil and platinum were used as the basic chemotherapy regimens, with or without targeted therapy, and no additional injection of PCSK9 inhibitors
  Interventions: Drug: standard advanced first-line regimen group
- PCSK9 inhibitor in combination with standard advanced first-line regimen group (Experimental): Fluorouracil and platinum as the base chemotherapy regimen, with or without targeted therapy, was administered subcutaneously at a fixed dose of 150 mg of PCSK9 inhibitor every two weeks starting on day 1 of patient enrollment
  Interventions: Drug: PCSK9 inhibitor in combination with standard advanced first-line regimen group

INTERVENTIONS:
Drug: PCSK9 inhibitor in combination with standard advanced first-line regimen group — Fluorouracil and platinum as the base chemotherapy regimen, with or without targeted therapy, was administered subcutaneously at a fixed dose of 150 mg of PCSK9 inhibitor every two weeks starting on day 1 of patient enrollment
  Arms: PCSK9 inhibitor in combination with standard advanced first-line regimen group
Drug: standard advanced first-line regimen group — Fluorouracil and platinum were used as the basic chemotherapy regimens, with or without targeted therapy, and no additional injection of PCSK9 inhibitors
  Arms: Late standard first-line treatment regimen group

SUMMARY:
The purpose of this study is to preliminarily observe the efficacy and safety of PCSK9 inhibitors in combination with standard advanced first-line regimens in the treatment of advanced colorectal cancer with pMMR/MSS.

DETAILED DESCRIPTION:
The purpose of this study is to preliminarily observe the efficacy and safety of PCSK9 inhibitors in combination with standard advanced first-line regimens in the treatment of advanced colorectal cancer with pMMR/MSS. To evaluate progression-free survival (PFS) after PCSK9 inhibitor combination, overall survival (OS) after PCSK9 inhibitor combination, and to evaluate the safety and tolerability of PCSK9 inhibitor combination therapy based on NCI-CTCAE version 4.03, and to further explore efficacy predictive biomarkers based on changes in the expression of specific immune markers in blood and tissue specimens at baseline and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited, and signed informed consent;
2. Histologically confirmed colorectal adenocarcinoma with pMMR/MSS;
3. Colorectal cancer with distant metastasis or inability to be radically surgically resected as assessed by imaging examination Patient;
4. Immunohistochemistry or sequencing to evaluate the high expression status of PCSK9 in tumors;
5. ECOG score 0-1;
6. Expected survival ≥ 3 months.

Exclusion Criteria:

1. Hypocholesterolemia, hypolipidemia and its family history, previous allergic reaction to PCSK9 inhibitors History of allergic reaction to PCSK9 inhibitors;
2. preoperative pathological diagnosis of advanced colorectal adenocarcinoma without pMMR/MSS, with the chance of radical surgical treatment;
3. Hypolipidemia caused by combination with other long-term lipid-lowering drugs;
4. malignancies other than colorectal cancer with negligible risk of metastasis or death (e.g., expected 5-year OS >90%) within 5 years prior to enrollment and for which a radical outcome is expected after treatment (e.g., adequately treated carcinoma in situ of the uterine cervix, basal or squamous cell skin cancers, limited prostate cancers treated for radical purposes, ductal carcinomas in situ treated for radical purposes surgically), with the exception of (b) the following;
5. history of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis;
6. major surgery within 4 weeks prior to enrollment or incomplete recovery from previous surgery;
7. systemic immunostimulatory drug therapy (including but not limited to interferon or IL-2) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to enrollment;
8. pre-existing or clinically significant CNS disease at screening, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndromes, or psychiatric disorders;
9. receipt of systemic corticosteroids (>10 mg/d prednisone equivalent) or other systemic immunosuppressants, etc. within 2 weeks prior to randomization;
10. previous allogeneic bone marrow transplantation or previous solid organ transplantation;
11. subjects who, in the judgment of the Investigator, have any factors affecting compliance with the protocol, including uncontrollable medical, psychological, familial, sociological, or geographic conditions; or who are unwilling or unable to comply with the procedures required in the study protocol;
12. history of idiopathic pulmonary fibrosis, drug-induced pneumonia, organic pneumonia (i.e., occlusive bronchiolitis), idiopathic pneumonia, or evidence of active pneumonia on CT scan of the chest at the time of screening; 13. receipt of any live vaccine (e.g., vaccines against infectious diseases such as influenza vaccine, varicella vaccine, etc.) within 4 weeks (28 days) prior to randomization

14. Pregnant or lactating female patients;

15. Hypersensitivity to fluorouracil-based or platinum-based agents or their excipients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2028-04-06 (Estimated); Study Completion 2028-05-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rateObjective response rate (ORR) | 5years
  Objective response rate (ORR) after PCSK9 inhibitor in combination with standard advanced first-line regimen in patients with advanced colorectal cancer with pMMR/MSS

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5years
  Progression-free survival (PFS) after PCSK9 inhibitor combination therapy
Overall survival (OS) | 5years
  Overall survival (OS) after PCSK9 inhibitor combination therapy

OTHER OUTCOMES:
Safety evaluation index | During the study
  According to NCI-CTCAE version 4.03, the safety and tolerability of PCSK9 inhibitor combination therapy

IPD SHARING:
Plan to Share IPD: No